CLINICAL TRIAL: NCT03918369
Title: A Multicenter Controlled Study of the Intracorporeal Mechanical Side-to-side Isoperistaltic Anastomosis Versus Extracorporeal Anastomosis in Laparoscopic Right Hemicolectomy: HEMI-D-TREND-study
Brief Title: Study of the Intracorporeal Versus Extracorporeal Anastomosis in Right Hemicolectomy: HEMI-D-TREND-study
Acronym: HEMI-D-TREND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Mireia Pascua-Solé (Unknown); Laura Mora-Lopez (Unknown); Anna Pallisera-Lloveras (Unknown); Sheila Serra-Pla (Unknown); Ricard Sales (Unknown); Beatriz Espina (Unknown); Luis Romangolo (Unknown); Anna Serracant (Unknown); Cristina Ruiz (Unknown); Mº José Mañas Gomez (Unknown); Angels Montserrat-Marti (Unknown); Mireia Merichal (Unknown); Carlos Cerdán-Santacruz (Unknown); Antonio Sanchez (Unknown); Helena Vallverdú (Unknown)
Responsible Party: Principal Investigator, Xavier Serra-Aracil, Head of Colorectal Unit, Corporacion Parc Tauli
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEMI-D-TREND-2019
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Colon Cancer
Keywords: Right Colon Cancer,; Right hemicolectomy; Laparoscopic right hemicolectomy; Intracorporeal anastomosis
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: A multicenter prospective, non-randomized, controlled study of the intracorporeal mechanical side-to-side isoperistaltic anastomosis versus extracorporeal anastomosis in laparoscopic right hemicolectomy. TREND-study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Intracorporeal anastomosis (Experimental): Laparoscopic right hemicolectomy with intracorporeal mechanical side-to-side isoperistaltic anastomosis.
  Interventions: Procedure: Laparoscopic right hemicolectomy with intracorporeal anastomosis.
- Laparoscopic extracorporeal anastomosis (Active Comparator): Laparoscopic right hemicolectomy with extracorporeal anastomosis.
  Interventions: Procedure: Laparoscopic right hemicolectomy with extracorporeal anastomosis.

INTERVENTIONS:
Procedure: Laparoscopic right hemicolectomy with intracorporeal anastomosis. — Intracorporeal anastomosis group The laparoscopic right hemicolectomy with intracorporeal mechanical side-to-side isoperistaltic anastomosis. In this procedure, intracorporeal division of the mesoileum and transverse colon is performed, as shown in the animation. The ileum and transverse colon are divided with the Endopath® Echelon Flex ™ 60 stapler. The specimen is inserted in a plastic bag. Side-to-side isoperistaltic mechanical anastomosis is performed using the same endostapler. A running suture is performed of the mechanical suture orifice, with another reinforcing suture with Monocryl ™ (poliglecaprone 25) or with STRATAFIX ™ Spiral Knotless barbed suture. The specimen is extracted through a Pfannestiel minilaparotomy (3.5-4 cm) Wound Protector
  Arms: Laparoscopic Intracorporeal anastomosis
Procedure: Laparoscopic right hemicolectomy with extracorporeal anastomosis. — Laparoscopic right hemicolectomy with extracorporeal anastomosis with the technical features of each center
  Arms: Laparoscopic extracorporeal anastomosis

SUMMARY:
INTRODUCTION: Colorectal cancer is the second most frequent cancer in the Western world. Roughly a third of colorectal tumors are located in the right colon, and right hemicolectomy surgery is the treatment of choice in non-disseminated right colon cancer and other benign pathologies. Despite the introduction of laparoscopy and multimodal fast-track perioperative management programs in recent years, postoperative complication rates remain high. The most serious complication is anastomotic leak (AL), which is associated with increased mortality, longer hospital stay, and reduced quality of life due to the presence of ostomies. For a long time, the importance of ileo-colic AL was underestimated. However, the ANACO study, conducted in 52 hospitals in our environment, reported a rate of AL of 8.4% with a range of 0 to 35%. This wide range is due to the differences in the surgical procedures and anastomoses used (the surgical approach may be open or laparoscopic, and the anastomosis may be manual or mechanical, with all its variations).

The results of intracorporeal laparoscopic anastomosis in the literature vary widely and, are discordant, although those reported so far estimate a DA less than 2%. But the latest publications report low rates of morbidity and of surgical space infection (SSI). The main problem with this technique is that it requires a learning curve somewhat greater than the others and its results depend on the skill of the surgeon and his casuistry. For all these reasons, it is necessary to carry out comparative studies that favor the use of this technique as gold standard.

The multicentre, controlled and randomized controlled studies have the disadvantage that randomization in centers not used with one of the techniques does include a learning curve bias. Besides the fact that in a center there is a belief that one of the techniques is superior to the other, it is not ethical to randomize the techniques. This situation has encouraged us to perform a non-randomized TREND-study design (Transparent Reporting of Evaluations with Non-randomized Designs-TREND).

Main objective:

To assess if laparoscopic right hemicolectomy, with anastomosis, obtains better results than laparoscopic with extracorporeal anastomosis and open surgery in terms of global morbidity, surgical space infection, anastomotic leak, re-interventions and hospital stay, in the first 30 postoperative days.

Secondary objectives:

To analyze the rate of anastomotic leak (AL) and organ-cavitary infections in each hospital.

* Compare the results obtained with those published in the literature.
* Try to identify the risk factors associated with AL.
* Analyze the comorbidities associated with the type of incision made for the extraction of the surgical piece, in intra and extracorporeal anastomosis

DETAILED DESCRIPTION:
Study Design: TREND-study design (Transparent Reporting of Evaluations with Non-randomized Designs-TREND):

A multicenter prospective, non-randomized, controlled study of the intracorporeal mechanical side-to-side isoperistaltic anastomosis versus extracorporeal anastomosis in laparoscopic right hemicolectomy. TREND-study.

Study procedure

Intracorporeal anastomosis group The laparoscopic right hemicolectomy with intracorporeal mechanical side-to-side isoperistaltic anastomosis. In this procedure, intracorporeal division of the mesoileum and transverse colon is performed, as shown in the animation. The ileum and transverse colon are divided with the Endopath® Echelon Flex ™ 60 stapler. The specimen is inserted in a plastic bag. Side-to-side isoperistaltic mechanical anastomosis is performed using the same endostapler. A running suture is performed of the mechanical suture orifice, with another reinforcing suture with Monocryl ™ (poliglecaprone 25) or with STRATAFIX ™ Spiral Knotless barbed suture. The specimen is extracted through a Pfannestiel minilaparotomy (3.5-4 cm) Wound Protector Extracorporeal anastomosis group according to the usual technique in each center.

Expected duration of subject participation; what is done and when: Duration of the study two years.

Population

Patients diagnosed with adenocarcinoma of the right colon up to the hepatic angle after complete colonoscopy, biopsy, and chest, abdominal and pelvic CT, and chest radiography, of the participating hospitals.

Recruitment Plan

Centers intracorporeal group: Parc Taulí University Hospital, Spain. Hospital Universitario Joan XXIII de Tarragona, Spain. Hospital de Cancer de Barretos. Brazil

Centers extracorporeal group: Consorcio Hospitalario de Terrassa (Barcelona), Spain. Hospital de Universitario de Vich (Barcelona), Spain. Hospital Universitario Arnau de Vilanova de Lleida, Spain. Hospital Santa Tecla de Tarragona, Spain. Hospital Universitario Sant Joan de Reus (Tarragona), Spain.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with right colon neoplasia non-metastatic.
* Indication of right hemicolectomy and ileo-colic anastomosis.
* Over 18 years.
* Scheduled surgery intervened by the team of surgeons of the Coloproctology Unit of each participating hospital.
* Patients who undergone a perioperative management program corresponding to the usual practice and technique of each hospital.

Exclusion Criteria:

* Colon neoplasms from other locations.
* T4 tumor stage and stage IV of the TNM classification.
* ASA IV (American Society Anesthesiologists).
* Non-optimal nutritional status (preoperative albumin ≤3.4 g / dl).
* Do not sign informed consent.
* Pregnant patients.
* Liver cirrhosis.
* Chronic renal insufficiency in dialysis treatment.
* BMI <18 and> 35 Kg / m

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Percentage of anastomotic leak (AL) | 30 days
  Percentage of anastomic leak (defined in accordance with Peel et al.).
Rate of global morbidity | 30 days
  Dindo-Clavien Classification
Rate of Surgical site infection | 30 days
  SSI in accordance with the Center for Disease Control (CDC) National Nosocomial Infection Monitoring System
Rate of Re-interventions | 30 days
  Percentage of re-interventions due to surgical complications

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Serra-Aracil, MD, PhD, Principal Investigator — Corporacio Parc Tauli. Parc Tauli University Hospital
Locations (1):
- Hospital Universitario Parc Tauli de Sabadell, Sabadell, Barcelona, Spain

REFERENCES:
- [Background] Frasson M, Granero-Castro P, Ramos Rodriguez JL, Flor-Lorente B, Braithwaite M, Marti Martinez E, Alvarez Perez JA, Codina Cazador A, Espi A, Garcia-Granero E; ANACO Study Group. Risk factors for anastomotic leak and postoperative morbidity and mortality after elective right colectomy for cancer: results from a prospective, multicentric study of 1102 patients. Int J Colorectal Dis. 2016 Jan;31(1):105-14. doi: 10.1007/s00384-015-2376-6. Epub 2015 Aug 28. PMID 26315015
- [Background] Frasson M, Flor-Lorente B, Rodriguez JL, Granero-Castro P, Hervas D, Alvarez Rico MA, Brao MJ, Sanchez Gonzalez JM, Garcia-Granero E; ANACO Study Group. Risk Factors for Anastomotic Leak After Colon Resection for Cancer: Multivariate Analysis and Nomogram From a Multicentric, Prospective, National Study With 3193 Patients. Ann Surg. 2015 Aug;262(2):321-30. doi: 10.1097/SLA.0000000000000973. PMID 25361221
- [Derived] Serra-Aracil X, Pascua-Sole M, Sanchez A, Gomez-Diaz CJ, Ruiz C, Espina B, Sierra JE, Lamas S, Vallverdu H, Corredera C, Veo C, Hoyuela C, Serracant A, Moreno F, Collera-Ormazabal P, Manas MJ, Merichal M, Cayetano-Paniagua L, Caro-Tarrago A; HEMI-D-TREND-study group. Intracorporeal vs extracorporeal anastomosis in laparoscopic right colectomy for colon cancer: a prospective multicenter cohort study (the Hemi-D-TREND study). Surg Endosc. 2025 Dec 1. doi: 10.1007/s00464-025-12401-0. Online ahead of print. PMID 41326726